CLINICAL TRIAL: NCT04532892
Title: Efficacy and Tolerance of a Specialized Nutraceutical for Pre-burnout - a Randomized, Double Blind Placebo Controlled Study
Brief Title: A Specialized Nutraceutical for Pre-burnout
Acronym: WELBI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Pasteur de Lille (Other)
Responsible Party: Principal Investigator, Jean-Michel Lecerf, MD in nutrition and endocrinology, Institut Pasteur de Lille
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2019-A02049-48
Record Dates: First submitted 2020-07-09; First posted 2020-08-31 (Actual); Last update posted 2022-12-08 (Actual); Status verified 2022-12

CONDITIONS: Burn Out; Psychological Disturbance
Keywords: Burnout; Dietary Supplement; Anxiety; Stress; Plants
MeSH Terms: conditions — Burnout, Psychological; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Monocentric, double-blind, randomized, placebo-controlled, 2-parallel arm study on outpatients
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: During the whole study, neither the investigators nor the subjects will be aware of the product they test. Every effort will be made to maintain the blind during the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Morning and night tablets with no active ingrédients. Morning and night tablets are different.
  Interventions: Dietary Supplement: Placebo Meta 18.06 Day and Placebo Meta 18.06 Night
- Dietary supplément (Experimental): Morning and night tablets with active ingrédients. Morning and night tablets are different.
  Interventions: Dietary Supplement: Meta 18.06 Day and Meta 18.06 Night

INTERVENTIONS:
Dietary Supplement: Meta 18.06 Day and Meta 18.06 Night — 5 visits after screening (V0-V4), including questionnaires (V0-V2-V4), salivary tests (V0 & V4) and calls for antistress advices and adverse events, concomitant medication reporting & compliance (V1 & V3)
  Arms: Dietary supplément
Dietary Supplement: Placebo Meta 18.06 Day and Placebo Meta 18.06 Night — 5 visits after screening (V0-V4), including questionnaires (V0-V2-V4), salivary tests (V0 & V4) and calls for antistress advices and adverse events, concomitant medication reporting & compliance (V1 & V3)
  Arms: Placebo

SUMMARY:
High demands, professional overload and emotional stress are well known negative influences on mental health. Chronic stress-related occupational diseases, especially Burnout, are becoming an important issue. Burnout can be defined as a negative affective state consisting of emotional exhaustion, cognitive weariness and physical fatigue, which is caused by chronic psychosocial stress.

Currently, there is no standard treatment for Burnout but different forms of psychological interventions are usually attempted. Also the administration of anxiolytics, antidepressants and sedatives only targets symptoms with a risk of addiction.

Recently, adaptogen plants have shown promising effects (e.g. Siberian Ginseng, Panax Ginseng, Rhodiola rosea and Ashwagandha) by increasing the body's ability to resist stress and exert a balancing effect on various systems of the body.

This study is focused on the effect of a specialized nutraceutical, containing adaptogen plants (Ashwagandha, Rhodiole rosea, Ginseng) as well as Vitamins and minerals (e.g. Vitamin C) needed for a normal hypothalamus-pituitary-adrenal (HPA) axis regulation in subjects suffering of early Burnout symptoms (pré-Burnout).

DETAILED DESCRIPTION:
High demands, professional overload and emotional stress are well known negative influences on mental health. Chronic stress-related occupational diseases, especially Burnout, are becoming an important issue. Burnout is an outcome of chronic depletion of the individual's coping resources resulting from prolonged exposure to stress, particularly work-related stress. In Germany, 8% of the working population believe they suffer from burnout syndrome. Among 7400 Czech Physicians, 34% feel they show symptoms and 83% perceive themselves at risk for having a burnout. Currently, the prevention of burnout has been discussed worldwide as absenteeism and other negative consequences related to job satisfaction, work performance and patient care lead to an economic burden.

Burnout can be defined as a negative affective state consisting of emotional exhaustion, cognitive weariness and physical fatigue, which is caused by chronic psychosocial stress. The 3 major dimensions of Burnout are emotional exhaustion, depersonalizations (cynicism) and a decreased sense of personal accomplishment or inefficacy. It is characterized by fatigue, mood disorder, sleep problems and cognitive impairment but is difficult to differentiate from depression as both illnesses are often related. The main difference with depression is at physiological level, mainly in Cortisol and dehydroepiandrosterone-sulphate (DHEA) levels.

Increased psychological stress affects the hypothalamus-pituitary-adrenal (HPA) axis regulation. During acute stress, plasma cortisol levels rise but during chronic stress, cortisol levels decline leading to a state of depletion. This depletion leads to a smaller increase of cortisol shortly after waking up, also known as the cortisol awakening response, leading to a disruption of the circadian rhythm, fatigue and a decreased mental performance. Next to cortisol, also DHEA levels are lower, especially in young Burnout patients. DHEA is an active hormone with effects on its own and a precursor of androgens and estrogens. It has a regenerative and protective role important for maintenance and restoration of health, thus very important in Burnout.

Next to hormones, also nutritional deficiencies related to HPA axis dysfunction could play a role in the development of Burnout. Vitamin C for example is needed for steroid biosynthesis, Niacin derivates are cofactors and Pantothenic acid and folic acid are vital to maintain steroid secretion from the adrenal cortex. Adrenocortical insufficiency has also been noted during biotin deficiency.

Diagnosis of Burnout often occurs via psychological scales (e.g. Maslach Burnout Inventory) with high scores for exhaustion and cynicism and low scores for professional efficacy.

Currently, there is no standard treatment for Burnout but different forms of psychological interventions are usually attempted. Also the administration of anxiolytics, antidepressants and sedatives only targets symptoms with a risk of addiction. Additionally, antidepressants lower also the cortisol levels putting Burnout patients even at higher risk of spiraling into Burnout.

Recently, adaptogens have also shown promising effects e.g. a clinical trial with Rhodiola rosea in 60 patients provided evidence of an antifatigue effect and an improvement in burnout symptoms. These botanicals (e.g. Siberian Ginseng, Panax Ginseng, Rhodiola rosea and Ashwagandha) are defined as substances that increase the body's ability to resist stress and exert a balancing effect on various systems of the body. These have shown to have an additive and beneficial effect in relieving HPA axis dysfunction in combination with vitamins and minerals and could thus have a beneficial effect in the treatment of Burnout.

This study is focused on the effect of a specialized nutraceutical, containing adaptogens (Ashwagandha, Rhodiole rosea, Ginseng) as well as Vitamins and minerals (e.g. Vitamin C) needed for a normal hypothalamus-pituitary-adrenal (HPA) axis regulation in subjects suffering of early Burnout symptoms (pré-Burnout).

ELIGIBILITY:
Inclusion Criteria:

* Female or male aged between 30 and 65 years (limits included),
* Presenting symptoms of stress, work or emotional overload based on :

  * COHEN questionnaire (score ≥ 21 allowed the inclusion),
  * CUNGI questionnaire (part 1: score ≥ 18 allowed the inclusion; part 2: score ≥ 30 allowed the inclusion).

Exclusion Criteria:

* Suffering from depression based on the Hospital anxiety and depression scale (depression score over 14),
* Considered in burn-out, based on MBI questionnaire:

  * Burnout > 30
  * Depersonalization > 12
  * Personnal achievement < 33 2 conditions should be fulfilling to exclude participant.
* Under nutritional supplement or drugs (psychotropics, betablockers) acting on mental health according to the investigator or stopped less than 3 months before the study.
* Diagnose of burn-out for less than 2y.

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2020-03-03 (Actual); Primary Completion 2022-11-25 (Actual); Study Completion 2022-11-25 (Actual)

PRIMARY OUTCOMES:
Mean score of the validated MQLI questionnaire (Multicultural Quality of Life Index) | 0 day (baseline), 60 days, 120 days
  A self-administered questionnaire. Score from 0 to 10 (from very bad Quality of Life to very good Quality of Life).

SECONDARY OUTCOMES:
Hospital Anxiety and depression questionnaire | 0 day (baseline) and 120 days
  A self-administered questionnaire:
  * A: Anxiety. A score over 7 describes an anxious behavior.
  * D: Depression. A score over 7 describes a depressive behavior.
Cungi questionnaire | 0 day (baseline) and 120 days
  This self-administered questionnaire is divided in two parts:
  * Part 1: stress factor scale. A score ≥ 18 is related to a high perception of environmental stress (many potential sources of stress).
  * Part 2: evaluation stress scale. Scores range from 11 to 66. A score ≥ 30 is related to an intermediate stress score.
Cohen questionnaire | 0 day (baseline) and 120 days
  This self-administered questionnaire contains 10 items. A score ≥ 27 corresponds to a high stress level.
MBI questionnaire (Maslach Burn Out Inventory Questionnaire) | 0 day (baseline) and 120 days
  This self-administered questionnaire will be filled by the subject at V0 and V4 visits.
  The questionnaire is subdivided in 3 categories:
  * Professional exhaustion,
  * Depersonalization,
  * Personal achievement.
  Each category will be analyzed as follow:
  Section A: Burnout
  * Total 17 or less: Low-level burnout
  * Total between 18 and 29 inclusive: Moderate burnout
  * Total over 30: High-level burnout
  Section B: Depersonalization
  * Total 5 or less: Low-level burnout
  * Total between 6 and 11 inclusive: Moderate burnout
  * Total of 12 and greater: High-level burnout
  Section C: Personal Achievement
  * Total 33 or less: High-level burnout
  * Total between 34 and 39 inclusive: Moderate burnout
  * Total greater than 40: Low-level burnout
PSQI Questionnaire (PITTSBURG SLEEP QUALITY INDEX) | 0 day (baseline) and 120 days
  The PSQI measured sleep quality and disturbances over a one-month interval across one global score and 7 component scores:
  * Duration of sleep (DURAT)
  * Sleep Disturbance (DISTB)
  * Sleep Latency (LATEN)
  * Day Dysfunction due to sleepiness (DAYDIS)
  * Sleep Efficiency (HSE)
  * Overall Sleep Quality (SLPQUAL)
  * Need Meds to Sleep (MEDS) The global score is calculated by the sum of the 7 subscores: DURAT + DISTB + LATEN + DAYDYS + HSE + SLPQUAL + MEDS.
SF-36 questionnaire | 0 day (baseline) and 120 days
  The SF36 measures health across 8 domains:
  * Physical function (PF);
  * Role physical (RP);
  * Bodily pain (BP);
  * General Health (GH);
  * Vitality (VT);
  * Social function (SF);
  * Role Emotional (RE);
  * Mental Health (MH).
  Two component summary measures can be calculated:
  * Physical Composite Score (PCS);
  * Mental Composite Score (MCS). One item considers the general health status (health transition, HT).
Saliva Cortisol | 0 day (baseline) and 120 days
  Saliva will be collected at the following time points at baseline (V0) and after 4 months of product consumption (V4) to analyze the salivary cortisol:
  * When the subject wakes up
  * 30 minutes after waking up
  * At 20 hours in the evening RIA method was used to analyze cortisol from saliva.

CONTACTS AND LOCATIONS:
Locations (1):
- NutrInvest - Institut Pasteur de Lille, Lille, Nord, France